CLINICAL TRIAL: NCT00999479
Title: Post Operative Continuous Active Combination Sex Steroids for the Prevention of Recurrent Endometrioma Formation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Endometrioma
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Norethindrone Acetate; ferrous fumarate; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monophasic OCP (Experimental): Patients randomized to this study arm will receive combined oral contraceptive pills. Patients will follow up at 2, 6, 12, 18 and 24 months. On follow up visits pts will have clinical assessment with vaginal and rectal examinations and with transvaginal ultrasonography. As a measure of compliance, patients will return their empty pill packages
  Interventions: Drug: Norethindrone acetate and ethinyl estradiol tablets, USP
- Placebo (Placebo Comparator): Patients assigned to this arm will use non-hormonal, barrier contraceptives to prevent pregnancy.Patients will follow up at 2, 6, 12, 18 and 24 months. On follow up visits pts will have clinical assessment with vaginal and rectal examinations and with transvaginal ultrasonography. As a measure of compliance, patients will return their empty pill packages.
  Interventions: Drug: ferrous fumarate (placebo) tablets

INTERVENTIONS:
Drug: Norethindrone acetate and ethinyl estradiol tablets, USP — Loestrin® 24 Fe provides a dosage regimen consisting of 24 white progestogen-estrogen contraceptive tablets and 4 brown ferrous fumarate (placebo) tablets.
  Each white tablet contains 1 mg norethindrone acetate and 20 mcg ethinyl estradiol. Each white tablet also contains the following inactive ingredients: acacia, lactose, magnesium stearate, starch, confectioner's sugar, and talc.
  Arms: Monophasic OCP
Drug: ferrous fumarate (placebo) tablets — Loestrin® 24 Fe provides a dosage regimen consisting of 24 white progestogen-estrogen contraceptive tablets and 4 brown ferrous fumarate (placebo) tablets. Each brown tablet contains ferrous fumarate, microcrystalline cellulose, magnesium stearate, povidone, sodium starch glycolate, and compressible sugar. The ferrous fumarate tablets do not serve any therapeutic purpose.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether or not continuous combined oral contraceptive pills (COCP's) decrease the risk of recurrent endometrioma formation. The investigators' hypothesis is that patients who have endometriomas surgically removed and then are started on COCP's will have a decreased incidence of recurrent endometrioma formation. The investigators' research protocol is designed to show a statistically significant decreased incidence of endometrioma formation in the hopes that physicians will use COCP's in patients they have removed an endometrioma in who do not desire immediate fertility. Long term, the investigators hope to establish a standard of care that COCP's be used postoperatively in appropriate candidates to decrease the chance of recurrent endometrioma formation.

DETAILED DESCRIPTION:
We plan to identify patients planning to undergo conservative surgery for endometrioma at the University of Oklahoma private practice OB/GYN clinic and at the University of Oklahoma Resident Women's clinic. After clear and appropriate consent and discussion regarding options, we plan to randomize patients to monophasic OCPs vs. placebo following surgery. We plan to enroll 35 patients in each arm and follow them for 24 months following the surgery. Surveillance with pelvic exam and transvaginal ultrasonography will occur at 2, 6 and 12 months. The patients surgery will be done prior to enrolling in our study. We will use information from their surgery only to confirm the diagnosis of endometrioma. The only procedure the subjects will undergo during the protocol are periodic transvaginal ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ovarian endometriotic cyst that has been surgically excited.

Exclusion Criteria:

* Current desire to achieve pregnancy or other contraindication to combined oral contraceptive pills.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine whether or not continuous combined oral contraceptive pills decrease the risk of recurrent endometrioma formation. | October 2011

SECONDARY OUTCOMES:
Long term, we hope to establish a standard of care that COCPs be used postoperatively in appropriate candidates to decrease the chance of recurrent endometrioma formation. | October 2011

CONTACTS AND LOCATIONS:
Overall Officials: Katie M Smith, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States